CLINICAL TRIAL: NCT02210858
Title: Phase I/II Study of Tipifarnib [Zarnestra, Farnesyltransferase Inhibitor R115777 (NSC 702818)] in Patients With Myeloproliferative Disorders
Brief Title: Tipifarnib in Treating Patients With Chronic Myeloid Leukemia, Chronic Myelomonocytic Leukemia, or Undifferentiated Myeloproliferative Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01606; NCI-2014-01606 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SUMC-NCI-38; NCI-38; CDR0000067864; CTEP 38 (Other: Stanford Cancer Institute); 38 (Other: CTEP); P30CA124435 (NIH); IRB-13343 (Other: Stanford IRB); NCT00005846 (obsolete NCT alias)
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Accelerated Phase of Disease; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Myelomonocytic Leukemia; Chronic Phase of Disease; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Recurrent Disease
MeSH Terms: conditions — Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Recurrence | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tipifarnib) (Experimental): Patients receive tipifarnib PO BID on days 1-21. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Tipifarnib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Tipifarnib — Given PO
  Other Names: R115777; Zarnestra

SUMMARY:
This phase 1-2 trial studies the side effects and how well tipifarnib works in treating patients with chronic myeloid leukemia, chronic myelomonocytic leukemia, or undifferentiated myeloproliferative disorders. Tipifarnib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To describe the toxicities of R115777 (tipifarnib) in adult patients with myeloproliferative disorders.
* To assess hematologic responses, including changes in white blood cell count and erythroid responses.

SECONDARY OBJECTIVES:

* To assess bone marrow cytogenetic responses to R115777.
* To analyze for the presence of neuroblastoma (N)/Kirsten rat sarcoma viral oncogene homolog (K-Ras) mutations in patient bone marrow samples.
* To analyze the effect of R115777 on Ras /DnaJ (Hsp40) homolog, subfamily A, member 1(HDJ-2) farnesylation in patient bone marrow/peripheral blood mononuclear cells.
* To analyze the effect of R115777 on mitogen-activated protein (MAP) kinase activation in patient bone marrow mononuclear cells.
* To perform colony forming unit granulocyte-macrophage (CFU-GM) cytotoxicity assays using patients' hematopoietic cells with R115777.

OUTLINE:

Patients receive tipifarnib orally (PO) twice daily (BID) on days 1-21. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a good hematologic response may continue treatment at the discretion of the treating physician.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with a diagnosis (> 3 months prior to enrollment) of:

  * Chronic myeloid leukemia (CML) (Philadelphia chromosome positive or polymerase chain reaction [PCR] positive for breakpoint cluster region [BCR]-Abelson murine leukemia viral oncogene homolog 1 [ABL]) in chronic phase with:

    * Persistent or progressive disease on maximum tolerated interferon therapy, or STI571 (if eligible and able to receive this drug), as evidenced by increasing white blood cell (WBC) count, peripheral blood myeloid immaturity and/or progressive anemia, and/or persistence or relapse of abnormal cytogenetic and/or molecular findings
    * Interferon or STI571 intolerant
  * CML (Philadelphia chromosome positive or PCR positive for BCR-ABL) in accelerated phase (< 20% blasts in the peripheral blood and bone marrow) with persistent or progressive disease on STI571 (if eligible and able to receive this drug)
  * CML patients are eligible if they have not received interferon or STI571 because they are allergic to these drugs or refuse their use
* Chronic myelomonocytic leukemia (CMML)

  * Proliferative-type (WBC > 12,000/mL)
  * Less than 5% blasts in the peripheral blood and < 20% blasts in the bone marrow
* Undifferentiated myeloproliferative disorder (UMPD)
* Atypical (i.e. Philadelphia chromosome-negative) CML
* Four weeks must have elapsed since the use of any previous pharmacotherapy including interferon, hematopoietic growth factors, and cytotoxic chemotherapy (6 weeks for prior mitomycin or nitrosoureas); hydroxyurea may be used to manage elevated cell counts in patients up to the time they begin investigational therapy
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patients are capable of swallowing capsules
* Total bilirubin is > 1.5 X the upper limit of normal (ULN) where the analysis is performed; for example, for Stanford University Hospital, the ULN for total bilirubin is 1.3
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) are > 2 X the ULN; for example, for Stanford University Hospital, the ULN for ALT is 35, and the ULN for AST is 41
* Serum creatinine of < 2.0
* Life expectancy > 4 months
* Written inform consent must be obtained

EXCLUSION CRITERIA:

* Blast crisis phase of CML and atypical CML/ undifferentiated myeloproliferative disorders
* Patients with > 20% blasts in the peripheral blood or bone marrow are excluded
* Prior allogeneic bone marrow transplantation
* Patients with severe disease other than CML, CMML, or UMPD which is expected to prevent compliance with the protocol
* Patients with septicemia or other severe infections
* Pregnant or breast-feeding females
* Women of reproductive age should use contraception while on study
* Patients may not receive androgens during the study
* Requirement for ongoing therapy with corticosteroids (> 10 mg/d prednisone or equivalent steroid dosage) other than as pre-medication for transfusions
* Patients with iron deficiency; if a marrow aspirate is not available, transferrin saturation must be > 20% and serum ferritin > 50 ng/mL; this exclusion criterion will be removed if the iron deficiency state is corrected before enrollment
* Patients with other contributing causes of anemia such as autoimmune or hereditary hemolytic disorders, gastrointestinal (GI) blood loss, B12 or folate deficiency, or hypothyroidism; patients who require platelet transfusions, or have thrombocytopenia-related bleeding
* Inability to return for follow-up visits/studies to assess toxicity and response to therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2000-05 (Actual); Primary Completion 2004-11-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Erythroid response in non-transfusion dependent patients | Up to 16 weeks
  Major response is defined as a > 2.0 g/dL rise in the hemoglobin after 2 to 4 cycles of therapy. Minor response is defined as a > 1.0 to < 2.0 g/dL rise in the hemoglobin after 2 to 4 cycles of therapy.
Erythroid response in transfusion-dependent patients | Up to 16 weeks
  Major response is defined as transfusion-independent after 2 to 4 cycles of therapy or a > 2.0 g/dL rise in hemoglobin without transfusion. Minor response is defined as > 1 to < 2.0 g/dL incremental rise in hemoglobin with a decrease in transfusion requirements of at least 50% compared to the mean transfusion requirement during the 8-week pre-study period.
Incidence of adverse events related to tipifarnib assessed by National Cancer Institute Common Toxicity version 2.0 | Up to 16 weeks
WBC response (complete response, defined as normalization of WBC count in patients with an elevated WBC count prior to treatment and partial response, defined as > 50% reduction in WBC count without normalization of WBC count) | Up to 16 weeks
  For all hematologic responses, the duration of response must be at least 2 months.

SECONDARY OUTCOMES:
Cytogenetic response (including Philadelphia chromosome-positive cells in metaphases in CML) | Up to 16 weeks
In vitro correlative studies (including N/K-Ras mutation analysis, N/K-Ras/HDJ-2 farnesylation, MAP kinase activation, and bone marrow CFU-GM cytotoxicity assays using tipifarnib with patients' hematopoietic cells) | Up to week 3 (course 4)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Greenberg, Principal Investigator — Stanford Cancer Institute
Locations (2):
- United States (2):
  - Stanford Cancer Institute, Palo Alto, California
  - University of Rochester, Rochester, New York